CLINICAL TRIAL: NCT06059885
Title: Tislelizumab Plus Tyrosine Kinase Inhibitor (TKI) as Adjuvant Therapy Versus Active Surveillance in Patients With HCC at High Risk of Recurrence After Curative Ablation: A Prospective Cohort Study
Brief Title: Tislelizumab Plus TKI as Adjuvant Therapy Versus Active Surveillance in Patients With HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, Fanping Meng, The Fifth Medical Centre of the General Hospital of PLA, Beijing 302 Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChiECRCT20210555
Record Dates: First submitted 2023-09-14; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Liver Neoplasms
Keywords: HCC; Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — tislelizumab; Tyrosine Kinase Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tislelizumab combined with tyrosine kinase inhibitor (TKI) treatment group (Experimental)
  Interventions: Drug: Tislelizumab plus tyrosine kinase inhibitor
- No-intervention group (No Intervention)

INTERVENTIONS:
Drug: Tislelizumab plus tyrosine kinase inhibitor — Lenvatinib, tyrosine kinase inhibitor (TKIs)
  Arms: Tislelizumab combined with tyrosine kinase inhibitor (TKI) treatment group

SUMMARY:
Background: Ablation is important radical treatment in hepatocellular carcinoma (HCC). However, the 5-year recurrence rate of HCC after ablation is up to 80%. Early and late recurrences are more likely related to tumor size, tumor multiplicity, vascular invasion, higher serum AFP level and disease etiology, etc. Some studies suggested that adjuvant immunotherapy might be associated with decreased recurrence and prolonged RFS. Adjuvant atezolizumab + bevacizumab (IMbrave 050) showed RFS improvement following curative resection or ablation. Currently, there is limited study on immunotherapy combined with TKI as postoperative adjuvant therapy for HCC. This is an open-label, prospective cohort study to compare the efficacy and safety of tislelizumab plus tyrosine kinase inhibitor (TKI) as adjuvant therapy versus active surveillance in HCC patients with high risk of recurrence after curative ablation.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients are ≥18 years, diagnosed with HCC confirmed by histopathology or cytology, with no prior targeted or immune checkpoint therapy for HCC, and have undergone curative ablation with no residual lesions according to imaging or pathological assessment. Patients are at high risk of recurrence meeting one of the following criteria:

solitary tumor >2cm but ≤5cm, or multiple tumors ≤4tumors and all≤5cm； poor tumor differentiation； macrovascular invasion of the portal vein(Vp1/Vp2) ； the absence or infiltration of a tumor capsule ； AFP≥32ng/ml； HBV DNA ≥105IU/ml； history of recurrence after curative treatment； family history of tumors.

Exclusion Criteria:

Concurrent with other primary malignant tumors; severe coagulation dysfunction or severe thrombocytopenic purpura; There is serious infection or organ failure; have previously received targeted drugs or other PD-1 antibody therapy;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Tumor recurrence rate (DRR) | 52 weeks
  Thoracic and abdominal enhanced MRI/CT and abdominal B-ultrasonography were performed before radical treatment, thoracic and abdominal enhanced MRI/CT and abdominal B-ultrasonography were performed after adjuvant treatment, and then thoracic and abdominal enhanced MRI/CT and abdominal B-ultrasonography were performed every 12 weeks. Tumor changes were evaluated by imaging. In addition, we will evaluate adverse events and death events: classify and grade adverse events, record the time and cause of death of patients. Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Fanping Meng, Principal Investigator — 302 Hospital Beijing, China
Locations (1):
- 302 Hospital, Beijing, Beijing Municipality, China